CLINICAL TRIAL: NCT03170050
Title: A Multicenter, Active-controlled, Randomized, Evaluator and Subject Blinded, Split-face, Comparative, Non-inferiority and Confirmatory Clinical Study of the Efficacy and Safety Between YYD701-2 and Restylane Perlane Lidocaine for Temporary Correction of Moderate to Severe Nasolabial Folds
Brief Title: Clinical Trial of YYD701-2 for Treatment of Nasolabial Folds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: YYP-YYD701_001
Record Dates: First submitted 2017-03-30; First posted 2017-05-30 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2017-12

CONDITIONS: Wrinkle Severity Rating Scale(WSRS) Grade 3 (Moderate) or 4 (Severe) of Nasolabial Folds
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: The Subjects are injected investigational devide(YYD701-2 or Restylane Perlane Lidocaine) in right or left nasolabial folds
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YYD701-2 (Experimental): YYD701-2 Hyaluronic Acid Gel and Lidocaine Hydrochlorid, total dose 1ml, single injection
  Interventions: Device: YYD701-2
- Restylane Perlane Lidocaine (Active Comparator): Restylane Perlane Lidocaine Hyaluronic Acid Gel and Lidocaine Hydrochlorid, total dose 1ml, single injection
  Interventions: Device: Restylane Perlane Lidocaine

INTERVENTIONS:
Device: YYD701-2 — HA Filler
  Arms: YYD701-2
Device: Restylane Perlane Lidocaine — HA Filler
  Arms: Restylane Perlane Lidocaine

SUMMARY:
A multicenter, active-controlled, randomized, evaluator and subject blinded, split-face, comparative, non-inferiority, Medical device Clinical trial.

This study is randomized, evaluator and subject blinded, split-face medical device Clinical trial. The Subjects are injected investigational device(YYD701-2 or Restylane Perlane Lidocaine) in right or left nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged between 30 and 75 years, inclusive
* Subjects who want improvement of nasolabial folds that are rated as grade 3 or 4 on Wrinkle severity rating scale(WSRS)
* Subjects who have visually symmetrical bilateral nasolabial folds
* Subjects who consent to discontinue all dermatological treatment or cure including wrinkle correction in and around infraorbital region during this trial
* Subjects who voluntarily decide to participate in this trial and provide written consent in the Informed Consent Form

Exclusion Criteria:

* Subject who have bleeding disorder in the past or present
* Other criteria as identified in the protocol

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
The change in Wrinkle Severity Rating Scale (WSRS) as evaluated by independent evaluator through Photographs. | from baseline to 24 weeks
  Score of WSRS assessed by the independent evaluator

SECONDARY OUTCOMES:
The change in Wrinkle Severity Rating Scale (WSRS) as evaluated by independent evaluator through Photographs. | from baseline to 2, 8, 16 weeks
  Score of WSRS assessed by the independent evaluator
The change in Wrinkle Severity Rating Scale (WSRS) as evaluated by investigator. | from baseline to 2, 8, 16, 24 weeks
  Score of WSRS assessed by the investigator
Proportion of subjects with a ≥ 1 point on Global Aesthetic Improvement Scale as evaluated by an investigator | 2, 8, 16, 24 weeks after week 0 (injection date)
  Score of GAIS assessed by the investigator
Proportion of subjects with a ≥ 1 point on Global Aesthetic Improvement Scale as evaluated by a subject | 2, 8, 16, 24 weeks after week 0 (injection date)
  Score of GAIS assessed by subject
Proportion of subjects with a ≥ 1 point change on Wrinkle Severity Rating Scale as evaluated by independent evaluator through Photographs. | from baseline to 2, 8, 16, 24 weeks
  Score of WSRS assessed by the independent evaluator
Proportion of subjects with a ≥ 1 point change on Wrinkle Severity Rating Scale as evaluated by the investigator | from baseline to 2, 8, 16, 24 weeks
  Score of WSRS assessed by the investigator
Visual Analogue Scale as evaluated by a subject | week 0 (injection date)
  Score of VAS assessed by subject

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Chung-Ang Univ. Medical Center, Seoul
  - Konkuk University Medical Center, Seoul